CLINICAL TRIAL: NCT05876143
Title: Ambispective Open Multicentric Study Evaluating Clinical Results of Unicondylar Knee Arthroplasty Performed With U-Knee/Uni-Kroma Implants
Brief Title: Ambispective Multicentric Study Evaluating UKA With U-Knee/Uni-Kroma Implants
Status: Recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-01
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Unicompartmental Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Fixed cementless UKP: Patient implanted with a fixed cementless Unicompartmental prosthesis
  Interventions: Device: Unicompartmental knee arthroplasty
- Fixed cemented UKP: Patient implanted with a fixed cemented Unicompartmental prosthesis
  Interventions: Device: Unicompartmental knee arthroplasty
- Mobile Cementless UKP: Patient implanted with a mobile cementless Unicompartmental prosthesis
  Interventions: Device: Unicompartmental knee arthroplasty
- Mobile Cemented UKP: Patient implanted with a mobile cemented Unicompartmental prosthesis
  Interventions: Device: Unicompartmental knee arthroplasty
- Fixed Cementless UKP (TIT coating): Patient implanted with a fixed cementless Unicompartmental prosthesis coating with "TIT"
  Interventions: Device: Unicompartmental knee arthroplasty

INTERVENTIONS:
Device: Unicompartmental knee arthroplasty — Knee joint could be subject to natural or pathological wear or shocks (primary or secondary evolutive or traumatic osteoarthritis) which cause pain and reduced mobility of the knee.
  When only one lateral or medial compartment of the femoro-tibial knee joint is affected, the treatment of unicompartmental femoro-tibial osteoarthritis of the knee is generally carried out by the implantation of a so-called unicondylar knee prosthesis (UKP), in order to reduce pain and improve joint mobility of the knee compared to the preoperative state.

SUMMARY:
This clinical investigation was led as a post-market clinical follow-up study (post-market device development stage).The main objective of this study is to collect short- and medium-term clinical data on the unicondylar knee prosthesis U-Knee / Uni-Kroma, in order to evaluate the performance of these implants.

ELIGIBILITY:
Inclusion Criteria:

- All patients using a U-Knee / Uni-Kroma unicompartmental knee prosthesis and benefiting from the social security affiliation scheme.

Exclusion Criteria:

* Patients who objected to participating in the study and the processing of their data
* Patients unable to understand the surgeon's instructions to complete their questionnaires or perform postoperative follow-up
* Patients who already have a unicompartmental prosthesis on the knee in question that need to be revised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adult for whom a unicondylar knee prosthesis is indicated according to U-Knee / Uni-Kroma instructions for use. Patients will be followed according to current practice
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 5 years
  Assess the survival rate of the investigational medical devices at 5 year follow-up

SECONDARY OUTCOMES:
Survival rate | 12-18 months to 10 years
  Assess the survival rate of the investigational medical devices at 12-18 months, 3 years and 10 years follow-up
Functional improvement | From pre-operative to 10 years
  Restoration of mobility and pain reduction evaluation using IKS score
Functional improvement | From pre-operative to 10 years
  Evaluate pain, symptoms, activities of daily life and sports activity using KOOS score
Forgetfulness of prosthesis | From pre-operative to 10 years
  Evaluate the degree of forgetfulness of the prostheses using FJS- score
Activity | From pre-operative to 10 years
  Evaluate the degree of activity using Devane score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Lyon Sud, Pierre-Bénite, France